CLINICAL TRIAL: NCT07209176
Title: A Clinical Trial to Address Physician- and Patient-based Barriers to NGS Testing
Brief Title: Physician- and Patient-based Barriers to NGS Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00505965; IRB00505965 (Other: JHM IRB)
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Prostate Cancer
Keywords: metastatic prostate cancer; next-generation sequencing
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider nudge and patient education at time of enrollment (Experimental): The provider level component (implemented for all patients) will be a "nudge" to physicians to order testing via a single email documenting their NGS testing rate relative to the Johns Hopkins top performer and, for those not in the top 20%, a link to the most recent American Society of Clinical Oncology (ASCO) guidelines recommending testing. In addition, there will be a patient component that is a one-page handout of educational material about NGS testing to be sent after their initial visit via email or mail.
  Interventions: Other: Provider-level and patient-level
- Provider component and patient education at end of study (Experimental): The provider level component (implemented for all patients) will be a "nudge" to physicians to order testing via a single email documenting their NGS testing rate relative to the Johns Hopkins top performer and, for those not in the top 20%, a link to the most recent ASCO guidelines recommending testing. The patient educational material will be provided by email or mail (if no email on file) to those who randomized to this arm.
  Interventions: Other: Provider-level and patient education at end of study

INTERVENTIONS:
Other: Provider-level and patient education at end of study — The provider level component will involve an email to each of the genitourinary medical oncologists at Johns Hopkins with their NGS testing rate from preliminary data and compare this rate to the mean. The initial email will also include the 2025 ASCO guideline recommending somatic testing in virtually all metastatic prostate cancer patients. Providers who do not have baseline NGS testing rates available will also be emailed. Providers will subsequently be emailed their updated NGS testing rate at the conclusion of the study period.
  Patients will also receive a one-page patient educational material (via email, or mail if no email on file) on advanced prostate cancer that includes education on somatic NGS testing at the end of the study period.
  Arms: Provider component and patient education at end of study
Other: Provider-level and patient-level — In addition to the provider component, patients will also receive a one-page patient educational material (via email, or mail if no email on file) on advanced prostate cancer that includes education on somatic NGS testing. The email will be sent by the MyChart Recruitment Innovation team. Those without email on file will have the same message and attachment sent via mail by our study coordinator.
  Arms: Provider nudge and patient education at time of enrollment

SUMMARY:
The goal of this study is to improve next-generation sequencing (NGS) testing rates at Johns Hopkins in patients with metastatic prostate cancer. Investigators believe by targeting two barriers, provider-level and patient-level, will improve the testing rate of NGS at Johns Hopkins.

DETAILED DESCRIPTION:
Next-generation sequencing is recommended by national guidelines in metastatic prostate cancer to inform prognosis, treatment decisions, and eligibility for clinical trials. However, rates are low nationally and around 50-60% at Johns Hopkins. Analysis found that older patients and patients who are not married are less likely to have testing performed. The goals and objectives of this proposed clinical trial are to improve NGS testing rates at Johns Hopkins using a multidisciplinary approach to improve the care of patients living with metastatic prostate cancer and reduce disparities. The hypothesis is that this initiative, which targets two barriers (provider-level and patient-level), will lead to higher rates of NGS ordering at Johns Hopkins.

ELIGIBILITY:
Inclusion Criteria:

* men diagnosed with metastatic prostate cancer
* seen by Johns Hopkins Medical Oncology as a new patient visit between January 1, 2025 and December 31, 2026

Exclusion Criteria:

- Patients who have already had NGS testing performed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-09-06 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Next-Generation Sequencing (NGS) testing by arm | 1 year

SECONDARY OUTCOMES:
Percentage of patients with sociodemographic and clinical characteristics who have had NGS testing compared to those without NGS testing during the study period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Marshall, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States